CLINICAL TRIAL: NCT06418399
Title: The Role of Central Sensitization in Pain, Functionality, and Quality of Life in Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 22.04.2024.354
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Central Sensitization
Keywords: Central Sensitization; cancer patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cancer patients — Patients aged between 18 and 80 years with cancer-related pain lasting for more than 3 months will be included.

SUMMARY:
Pain is one of the most important and challenging symptoms in cancer patients. Depending on the stage of cancer, approximately 40% to 70% of patients complain of pain. With the increasing lifespan of cancer patients due to developing treatments, pain palliation has become even more crucial to improve their quality of life. Cancer-related pain can develop through multiple mechanisms such as the tumor itself, metastasis, or the methods used in treatment. The type of pain can be nociceptive, neuropathic, or mixed.

Central sensitization refers to the increased response of central nervous system nociceptive neurons to normal or subthreshold stimuli. Recently, central sensitization (CS) has been recognized as a potential pathophysiological mechanism underlying a group of chronic pain diseases such as fibromyalgia, temporomandibular joint disorder, irritable bowel syndrome, interstitial cystitis, tension-type headache, and chronic low back pain. Since pain perception varies from person to person, physicians should assess the character of pain thoroughly and not rely solely on peripheral pain treatment in cases with a component of central sensitization. The lack of evaluation of the extent to which central sensitization affects patients and the failure to fully determine the factors influencing it appear to be clinical limitations for now.

There are studies suggesting that central sensitization may be a significant factor in chronic refractory pain in cancer patients, indicating the need for consideration of alternative options to classical treatments. To the best of our knowledge, no study has been conducted in Turkey to investigate the frequency of central sensitization and its impact on treatment outcomes in chronic cancer pain patients visiting outpatient clinics. The aim of this study is to investigate the frequency of central sensitization and its effect on pain and quality of life in chronic cancer pain patients attending algology clinics in multiple centers in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years

  1. Diagnosis of cancer confirmed pathologically
  2. Experiencing cancer or cancer treatment-related pain complaints for more than 3 months

Exclusion Criteria:

* 1.Patients with chronic pain not related to cancer will be excluded from the study 2.Patients who do not provide consent to participate in the study 3.Patients with conditions such as dementia, traumatic brain injury, advanced psychiatric disorders (schizophrenia, etc.), chromosomal disorders (Down syndrome), genetic diseases (fragile X syndrome), and neurodegenerative diseases that may lead to mental disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 80 years with cancer-related pain lasting for more than 3 months will be included.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of central sensitization in cancer patients can be determined. | 1 year
  Central sensitization is a common condition in cancer patients and has negative consequences on pain, functionality, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Savaş Şencan, Assoc. Prof., Study Director — Marmara University Faculty of Medicine, Department of Pain Medicine; Serdar Kokar, Assoc. Prof., Study Director — Marmara University Faculty of Medicine, Department of Pain Medicine

IPD SHARING:
Plan to Share IPD: Undecided
The study is planned as multicenter, and data transfer will be conducted with other centers.

REFERENCES:
- [Background] Bouhassira D, Luporsi E, Krakowski I. Prevalence and incidence of chronic pain with or without neuropathic characteristics in patients with cancer. Pain. 2017 Jun;158(6):1118-1125. doi: 10.1097/j.pain.0000000000000895. PMID 28267066
- [Background] Petersel DL, Dror V, Cheung R. Central amplification and fibromyalgia: disorder of pain processing. J Neurosci Res. 2011 Jan;89(1):29-34. doi: 10.1002/jnr.22512. PMID 20936697
- [Background] Smart KM, Blake C, Staines A, Thacker M, Doody C. Mechanisms-based classifications of musculoskeletal pain: part 1 of 3: symptoms and signs of central sensitisation in patients with low back (+/- leg) pain. Man Ther. 2012 Aug;17(4):336-44. doi: 10.1016/j.math.2012.03.013. Epub 2012 Apr 23. PMID 22534654
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Nishigami T, Manfuku M, Lahousse A. Central Sensitization in Cancer Survivors and Its Clinical Implications: State of the Art. J Clin Med. 2023 Jul 11;12(14):4606. doi: 10.3390/jcm12144606. PMID 37510721